CLINICAL TRIAL: NCT00176306
Title: Levofloxacin Pharmacokinetics in the Severely Obese
Brief Title: Levofloxacin Pharmacokinetics (PK) in the Severely Obese
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Joel Thompson, PhD (Other)
Collaborators: Ortho-McNeil Pharmaceutical (Industry)
Responsible Party: Sponsor-Investigator, Joel Thompson, PhD, PhD, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAPSS-391; CAPSS-391 (Other: Johnson & Johnson)
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2012-10-12 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Obesity; Critical Illness
MeSH Terms: conditions — Obesity; Critical Illness | interventions — Levofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levofloxacin (Experimental): Patients receiving levofloxacin 750mg IV
  Interventions: Drug: Levofloxacin 750 mg IV

INTERVENTIONS:
Drug: Levofloxacin 750 mg IV — PK in obesity
  Other Names: Levaquin

SUMMARY:
Obesity is known to affect the concentrations of certain medications in the body. Levofloxacin is a commonly used antibiotic. Based on what the investigators know about levofloxacin and how it moves through the body, obesity may affect levofloxacin concentrations. This study aims to show the effect of obesity on levofloxacin concentrations.

The hypothesis is as follows: A 750 mg intravenous (IV) dose of levofloxacin administered to severely obese, critically ill patients will yield serum concentrations that are likely to be therapeutic.

DETAILED DESCRIPTION:
Although the pharmacokinetics of levofloxacin have been consistent in various study populations, obese and critically ill individuals are likely to demonstrate altered distribution and clearance of levofloxacin, in addition to potentially having altered serum concentrations. Thus, the following study proposes to address the question: What are the effects of the combination of critical illness and severe obesity on the pharmacokinetics of levofloxacin. The data from this investigation will also be combined with obese ambulatory volunteer data to more accurately define the effects of obesity on the pharmacokinetic parameters of levofloxacin.

There are no comparisons in this study. The specific aims are:

1. Characterize pharmacokinetic parameters of levofloxacin in obese critically ill individuals: Cmax, Tmax, area under the concentration-time curve (AUC), volume of distribution, elimination rate, serum half-life, and urine clearance.
2. Determine the percentage of patients that achieve an AUC/MIC ratio* of 88, which is achieved in 72% of non-obese, non-critically ill patients and is correlated with efficacy.

Hospitalized subjects will be identified by medical or pharmacy house staff officers providing care in the intensive care unit and through computerized medication profiles provided by UKCMC or UTMB Pharmacy Services. Once an investigator determines eligibility, a recommendation will be made to enroll the patient in the study to the attending physician.

After obtaining permission to enroll the subject, the investigator will obtain informed consent from the patient or his/her appropriate surrogate. The decision of competence will be made by the physician, in conjunction with family members, if available. Assessment of competence for providing informed consent will be documented in the medical record via the statement below:

"The patient was fully assessed and is/is not competent to agree to the study. Family members, including the patient's surrogate, were present for the assessment and agree the patient is/is not competent for purposes of study entry. This assessment and conversation with the family was witnessed by nurse assigned to the patient's care."

The informed consent document will be signed and an original copy will be placed in the patient's medical record. No study related orders will be written until the signed consent form is included in the medical record.

Ambulatory subjects will be identified by medical staff. Participants are likely to be recruited from physician clinics such as sleep clinic.

Research Procedures:

Ambulatory volunteers will be admitted for 24 hours to the UTMB or UK General Clinical Research Center. Hospitalized participants will be admitted to the UKCMC or UTMB hospital for reasons other than participation in the study. Each participant will receive a 750 mg intravenous levofloxacin dose.

A peripheral intravenous catheter will be placed in each arm for drug administration and serial blood sampling. Pre-existing intravenous access will be utilized when possible. Baseline serum chemistry and complete blood count will be obtained for each individual prior to the levofloxacin dose for screening purposes. Subjects will rest in a supine position while receiving a 750 mg intravenous dose of levofloxacin over 90 minutes. Serial blood samples will be obtained 1.5, 3, 4, 5, 8, 12, and 24 hours after the beginning of administration of levofloxacin. Urine collection will also be completed during the 24 hour study period.

Venous blood samples will be collected in 10 ml standard red-top vacuum tubes. The samples will be centrifuged for 10-15 minutes at 5000 rpm, the serum removed, and placed in a plastic vial suitable for freezing. The samples will be placed in a -80oC freezer until ready for shipment to the site for assay. Urine will also be collected during the 24 hour study period to assess renal function as well as measure drug elimination. Two aliquots will be extracted from the total urine volume: one for levofloxacin assay (storage procedure as above) and one for urine creatinine measurement (for 24 hour creatinine clearance). Urine aliquots and serum samples will be transported to the University of Kentucky College of Pharmacy for levofloxacin assay.

Ambulatory participants at the University of Texas Medical Branch will undergo a whole body potassium-40 counter scan in order to determine the percentage of adipose and lean body mass. This will consist of subjects lying in a supine position for 30 to 45 minutes under the whole body counter that is housed in the General Clinical Research Center at the University of Texas Medical Branch. The ambulatory volunteers will be scanned during the 24 hour study period.

Initial data to be collected include: age, height, weight, admitting diagnosis, serum creatinine, blood urea nitrogen, fluid intake/output, concomitant medications, concomitant disease states that might affect pharmacokinetics, any operating room procedures, documented or suspected infection site, pertinent microbiological culture results, and adverse drug reactions. Levofloxacin pharmacokinetics will be analyzed assuming a two-compartment model with first order elimination using WinNonLin 4.01 (Pharsight Corp, Mountainview, CA). Patients will be followed for 24 hours.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 55 years of age
2. Body mass index > 35 kg/m2
3. Has been prescribed levofloxacin, but the medication has not yet been administered (hospitalized cohort only)

Exclusion Criteria:

1. Hypersensitivity to fluoroquinolones
2. Creatinine clearance < 50 ml/min
3. Administration of levofloxacin within the previous 7 days
4. Pregnant or lactating females
5. Participation in another investigational protocol within the past 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2005-01; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard S Morehead, MD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Levofloxacin Arm: Patients receive commercially available levofloxacin 750mg solution for intravnous use
Period: Overall Study
Arm/Group | Levofloxacin Arm
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Levofloxacin Arm: patients receiving levofloxacin
Arm/Group | Levofloxacin Arm
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.4 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 15

OUTCOME MEASURES:

1. Primary Outcome: Plasma Concentration of Levofloxacin
Description: A peripheral intravenous catheter will be placed in each arm for drug administration and serial blood sampling. Pre-existing intravenous access will be utilized when possible. Subjects will rest in a supine position while receiving a 750 mg intravenous dose of levofloxacin over 90 minutes. Serial blood samples will be obtained 1.5, 3, 4, 5, 8, 12, and 24 hours after the beginning of administration of levofloxacin. Data will be presented as mean area under the curve +/- standard deviation.
Time Frame: 24 hours
Population: pilot study
Measure: Mean (Standard Deviation); unit: mg/L*hr
Groups:
- Levofloxacin Arm: Subjects receiving levofloxacin
Arm/Group | Levofloxacin Arm
Number analyzed (Participants) | 15
mg/L*hr | 76 (32)

ADVERSE EVENTS:
Time Frame: During infusion and study period
Arm/Group | Levofloxacin Arm
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

LIMITATIONS AND CAVEATS:
The number of ambulatory volunteers was low The acutely ill cohort was a heterogeneous population We remain unable to predict the precise effect of all of these different physiologic processes on drug pharmacokinetics

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No